CLINICAL TRIAL: NCT01466426
Title: The Role of FDG-PET/CT Imaging in the Management of Patients With Thromboembolic Disorders
Brief Title: The Role of FDG-PET/CT Imaging in the Management of Patients With Thromboembolic Disorders (The PETVET Study)
Acronym: PETVET
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Søren Hess, MD, MD, Odense University Hospital
Other Study IDs: NMA projekt K 59 PETVET
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Venous Thromboembolic Disease
Keywords: Venous thromboembolic disease; Deep veinous thrombosis; Pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- DVT confirmed
- DVT ruled out
- PE confirmed
- PE ruled out

SUMMARY:
This pilot study aims at validating 18F-flourodeoxyglucose positron emission tomography/computed tomography (FDG-PET/CT) in the detection and characterization of venous thromboembolism (VTE) in the entire human body, especially deep venous thrombosis (DVT) and pulmonary embolism (PE). On completion of this study the investigators will hopefully be able to demonstrate the importance of functional/molecular imaging technique in managing patients with this common and potentially fatal disorder.

DETAILED DESCRIPTION:
Acute DVT and PE are common and serious conditions. Highly effective treatment (most often anticoagulant agents) is available for acute VTE, but it is associated with potentially dangerous side effects. In addition, DVT and PE are just two manifestations of VTE, which can occur everywhere in the human organism. An underlying disease (i.e. cancer) is often a key factor in developing VTE.

Commonly used diagnostic imaging techniques in DVT and PE have a fair diagnostic accuracy, but do not address other important aspects of the disease. In contrast to this, FDG-PET/CT has the potential to contribute in VTE diagnosis by

* Differentiate between acute and chronic VTE
* Screening of the entire body for VTE (e.g. the pelvis where normal imaging techniques fail)
* Early diagnosis of underlying disease (e.g. cancer, with the possibility of early treatment)

This is a pilot study with the above mentioned objectives, and is part of a larger study addressing other aspects of FDG-PET/CT in VTE.

The investigators believe that their hypothesis that FDG-PET/CT imaging may introduce a new approach for detecting thrombi anywhere in the body, particularly in the venous system including the pelvis and the calves, will add a new dimension in treating patients with suspected PE. This technology will only detect acute thrombi and not chronic thrombi that no longer have activity, which will obviate unnecessary treatment in this population.

ELIGIBILITY:
Inclusion Criteria:

* Positive or negative diagnosis of VTE (DVT/PE)
* Age ≥ 50 years
* Informed consent obtained
* Symptoms < 1 week

Exclusion Criteria:

* Pregnant or lactating women
* Foreign language patients with a need for an interpreter
* Previous DVT or PE
* Known malignancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises the following patient groups: 10 patients with a positive diagnosis of DVT, 10 patients where clinically suspected DVT was ruled out, 10 patients with a positive diagnosis of PE, and 10 patients where clinically suspected PE was ruled out.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Proof-of-concept | During diagnostic workup
  Simple assessment of scans - positive or negative in the relevant patient categories

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Hess, MD, Study Chair — Odense University Hospital; Poul Henning Madsen, MD, Study Chair — Odense University Hospital
Locations (3):
- Denmark (3):
  - Dept. of Acute Medicine, Odense University Hospital, Odense
  - Dept. of Nuclear Medicine, Odense University Hospital, Odense
  - Dept. of Respiratory Medicine, Odense University Hospital,, Odense